CLINICAL TRIAL: NCT02606409
Title: Dexmedetomidine Versus Propofol for Prolonged Sedation in Poly Traumatized Mechanically Ventilated Patients
Acronym: DEXsedation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, MD, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/1548
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-06

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine intravenous sedation at 0.2-0.7 µg/kg/h for >24h.
  Interventions: Drug: Dexmedetomidine
- Propofol (Active Comparator): Propofol sedation at 10-70µg/kg/h for >24h.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine sedation at a starting dose of 0.2-7.0 µg/kg/hour.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Propofol — Propofol sedation at a starting dose of 10-70 µg/kg/hour.
  Other Names: Deprivan
  Arms: Propofol

SUMMARY:
Dexmedetomidine, a central and peripheral α2-receptor agonist distinct from GABA receptor for benzodiazepines and propofol, has been approved by the US Food and Drug Administration only for use up to 24 h in mechanically ventilated patients. The investigators aim to compare dexmedetomidine with propofol for sedation >24h in poly traumatized mechanically ventilated patients.

DETAILED DESCRIPTION:
The importance of optimizing the levels of sedation in critical care has been increasingly recognized. Many intensive care experts are focusing on maintaining a targeted ''ideal'' sedation level according to the individual patient's condition to avoid adverse events such as prolonged mechanical ventilation, respiratory depression, pneumonia, delirium, psychological problems, and increased treatment costs resulting from over sedation. Dexmedetomidine is a selective alpha-2-adrenoceptor agonist. It exerts both sedative and analgesic effects via mechanisms different from other sedatives such as midazolam and propofol, and provides sedation characterized by prompt response to stimuli with no respiratory depression. The investigators aim to compare dexmedetomidine with propofol for sedation >24h in poly traumatized mechanically ventilated patients. The investigators will perform a prospective, single center trial to investigate the safety and efficacy of dexmedetomidine for long-term sedation in poly traumatized mechanically ventilated ICU patients, in comparison with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheal Intubation
* Mechanical ventilation
* Poly traumatized
* ICU patients and estimated duration of sedation>24 h.

Exclusion Criteria:

* Patients with serious trauma in the central nervous system,
* with bleeding probably requiring surgical hemostasis,
* drug overdose within the last 30 days before study entry,
* pregnancy/lactation,
* contraindication to alpha-2-adrenoceptor agonists or antagonists,
* cardiovascular disease,
* conduction disturbances or difficulty in data collection or completing the study protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
percentage of time with in the target sedation range of Richmond Agitation Sedation Scale-3-0 | 3 days
  sedation goal is to maintain Richmond Agitation Sedation Scale from -3 up to 0

SECONDARY OUTCOMES:
serum BUN | 3-days
  Assessment of the serum level of BUN.
Serum creatinine. | 3-days
  Assessment of the serum level of creatinine.
Systolic blood pressure | 3- days.
  systolic blood pressure is measured every hour for 3- days.
diastolic blood pressure | 3- days.
  diastolic blood pressure is measured every hour for 3- days.
heart rate | 3- days.
  heart rate is recorded every hour for 3-days.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in Anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No